CLINICAL TRIAL: NCT01227798
Title: A Pilot Study to Evaluate the Safety and Efficacy of IFN-alfacon1 (INFERGEN) in the Treatment of Hospitalized Patients Presenting With Influenza-like Illnesses Due to the Pandemic 2009 Swine Origin Influenza A Virus (S-OIV) H1N1 and Other Circulating Influenza Viruses
Brief Title: Safety and Efficacy Study of Interferon to Treat Patients Hospitalized for Influenza
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dante Morra, MD, University Health Network
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-H1N1; 09-0599-B (Other: UHN Research Ethics Board)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-08

CONDITIONS: Influenza
Keywords: influenza A, H1N1
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — interferon alfacon-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 100 mM sodium Chloride and 25 mM sodium phosphate at pH 7.0 +/- 0.2
  Interventions: Drug: Placebo
- Infergen (Active Comparator): 15mcg subcutaneous injection at fill volume of 0.5mL
  Interventions: Drug: Interferon alfacon-1

INTERVENTIONS:
Drug: Interferon alfacon-1 — 15 mcg at fill volume of 0.5mL
  Other Names: Infergen
  Arms: Infergen
Drug: Placebo — Normal Saline
  Other Names: NS
  Arms: Placebo

SUMMARY:
A Pilot Study to Evaluate the Safety and Efficacy of interferon-Alfacon1 (INFERGEN) in the treatment of patients hospitalized with Influenza-like illness caused by a novel swine origin Influenza virus and other circulating Influenza Viruses.

The use of Interferon-alfacon1 as a co-treatment along with the standard of care antiviral is hypothesized to be safe. Clinical improvement of patients is hypothesized to be quicker.

DETAILED DESCRIPTION:
The purpose of this study is to see if using a medication called INFERGEN, can help get rid of the virus and/or can help the immune response to prevent the illness from getting worse in the lungs. We hope that INFERGEN will either prevent patients from getting worse and requiring intensive care or will decrease the time for which they will need intensive care.

The Interferon-alpha (also called Interferon-alphacon1 or IFN-alphacon1 or INFERGEN) is an immune molecule, which has been shown to work against different viruses (anti-viral). Interferon is the standard of treatment for patients with chronic (infection that has been there for a long time) hepatitis C (a virus which affects the liver over many years) by giving it for 6-12 months. It has also been used for a shorter time of up to 14 days, in a small study for patients with respiratory disease caused by SARS and seemed to help these patients get better more rapidly. It also has been shown to stop different Influenza viruses from growing in test tubes and in lung tissue. It has also been shown to decrease the immune response to prevent it from over-reacting to viruses.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Aged >=18 and < 70
* Hospitalized
* suspect, probable, confirmed influenza A
* symptom onset <8 days
* able to attend all scheduled visits

Exclusion Criteria:

* known hypersensitivity to interferon preparation
* pregnancy
* chronic liver disease
* moderate to severe congestive heart failure, grade III or IV left ventricular function
* previous history of serious psychiatric illness
* history of severe or active autoimmune disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of Clinically Important (moderate or severe) and serious adverse events | Up to two-months post-treatment
  occurrence, severity, time to onset, duration (number of days), seriousness, nature.

SECONDARY OUTCOMES:
Virologic Clearance | Day 1,2-4,7,10,14, (21)
  Clearance and/or reduction in copies/mL of viral RNA as determined by PCR and/or quantitative real-time PCR in respiratory secretions (nasopharyngeal swab, throat swab, sputum, ETT aspirate BAL)
Cytokines and PBMC | Day 1,2-4,7,10,14
  levels of pro-inflammatory cytokines in serum.
Clinical Improvement | Duration of hospitalization
  SOFA, LIS scores at baseline, 48hrs, 96hrs, day7. Days to defervesce, days of O2 requirement, days of cough, days hospitalized, days in ICU, days with ventilatory support, days on PEEP >10cm H2O.
  Death all causes 28 days, Death all causes duration of study.

CONTACTS AND LOCATIONS:
Overall Officials: Dante Morra, MD, MBA, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada